CLINICAL TRIAL: NCT05575596
Title: Impact Des inégalités Socio-économiques et Territoriales Sur la qualité de Vie pré et Post opératoire Des Scolioses Idiopathiques Prisent en Charge en Milieu pédiatrique
Brief Title: Influence of Social Deprivation and Remoteness on Quality of Life in Adolescent's Surgical Scoliosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Collaborators: Hôpital Necker-Enfants Malades (Other); Hopital Universitaire Robert-Debre (Other); Amiens University Hospital (Other); University Hospital, Rouen (Other); University Hospital, Lille (Other)
Responsible Party: Principal Investigator, Nathan DOLET, MD, University Hospital, Caen
Other Study IDs: ISASE001
Record Dates: First submitted 2022-10-03; First posted 2022-10-12 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Idiopathic Scoliosis
Keywords: inequality; remoteness; socio economic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The incidence of idiopathic scoliosis is 3% or approximatively 300,000 new cases per year in France. It is estimated that between 0.1 and 0.3% of patients will eventually require surgical management, between 500 and 1000 scoliosis are operated per year in France. To our knowledge, the impact of socio-economic and territorial inequalities on the quality of life before and after surgery of idiopathic scoliosis has not been studied previously.

Main objective:

-Assess the impact of socio-economic and territorial inequalities on the pre- and post-operative quality of life at 1 year after surgical idiopathic scoliosis management, in a French pediatric surgery multicenter cohort.

Secondary objective:

* Assess the impact of socio-economic and territorial inequalities on the quality of life pre and postoperative at 3 months after surgery on a French multicenter cohort.
* To assess the impact of severity and type of scoliosis on pre- and post-operative quality of life at 3 months and 1 year after surgery on a French multicenter cohort.

ELIGIBILITY:
Inclusion Criteria:

* Operated by posterior vertebral arthrodesis
* Opereted in pediatric surgery center
* Idiopathic scoliosis treated by surgery

Exclusion Criteria:

* Refusal to participate
* People unable to read or speak French (the questionnaire being in French)
* Non-idiopathic scoliosis

Ages: 10 Years to 25 Years | Sex: All
Age Groups: Child, Adult
Study Population: All patients operated in one of the participating pediatric surgery center (Paris centers : NECKER and Robert DEBRE, University Hospital of Caen, University Hospital of Amiens, University Hospital of ROUEN, University Hospital of LILLE). Only the patient operated by posterior vertebral arthrodesis will be included.
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2022-11-14 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Change from baseline quality of life (SRS-22) at one year after surgery depending on the socio-economic level and remoteness. | At 1 years after surgery. Baseline questionnaire will be assessed just before the surgery
  We will use the SRS-22 questionnaire, a specific questionnaire validated in French to assess the quality of life of patients with scoliosis.
  The questionnaire coverts different part of socio-economic levels including the salary, the educational level, the type of social security coverage, the parents' family situation (single parent, two-parent, blended couple) and the number of people and pieces in the habitation.
  The remoteness will be evaluated by the distance between the medical referent center and the habitation.

SECONDARY OUTCOMES:
Radiological data: angulation parameters | at the time of surgery and at one year fater surgery
  Scoliosis radiological parameters before and after surgery (just after and at 1 year after surgery) cobb, kyphosis, lordosis, pelvic incidence (unit of measure: angulation in degrees)
Radiological data : type of scoliosis | at the time of surgery and at one year fater surgery
  Scoliosis radiological parameters before and after surgery (just after and at 1 year after surgery): type of scoliosis (lenkee classification)
Clinical data: age | at the surgery
  Age at diagnosis and at surgery in months
Clinical data: weight | at the surgery
  weight (in kilograms)
Clinical data: previous treatments | at the surgery
  previous treatment for scoliosis (yes or no)
Clinical data: family history | at the surgery
  history of scoliosis in the family (yes or no)
Surgery data | during the firts year after the surgery
  Type of instrumentation, level of instrumentation, surgical complications (neurological, infectious).

CONTACTS AND LOCATIONS:
Locations (1):
- DOLET Nathan, Caen, Calvados, France

IPD SHARING:
Plan to Share IPD: Undecided